CLINICAL TRIAL: NCT04941235
Title: The Effectiveness of Different Techniques of Interscalene Brachial Plexus Block With General Anesthesia for Shoulder Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shery Shehata Kyriacos, Assistant Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 219:7/2019
Record Dates: First submitted 2021-06-20; First posted 2021-06-28 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Shoulder and Upper Arm Injury
Keywords: shoulder arthroscopy
MeSH Terms: conditions — Arm Injuries | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NU group (Active Comparator): Bth nerve stimulator and ultrasound guided interscalene brachial plexus block
  Interventions: Device: ultrasound and nerve stimulator
- U group (Active Comparator): Ultrasound guided interscalene brachial plexus block
  Interventions: Device: ultrasound and nerve stimulator
- N group (Active Comparator): Nerve stimulator guided interscalene brachial plexus block
  Interventions: Device: ultrasound and nerve stimulator
- C group (No Intervention): No block only IV analgesics

INTERVENTIONS:
Device: ultrasound and nerve stimulator — nerve stimulator and ultrasound guided interscalene brachial plexus block
  Arms: N group; NU group; U group

SUMMARY:
There are different techniques of interscalene brachial plexus block, we aimed to evaluate the effectiveness of 3 of them as analgesia during shoulder arthroscopy surgery under general anesthesia.

DETAILED DESCRIPTION:
Prospective randomized controlled study

There were 4 groups included in our study:

Group N: nerve stimulator guided interscalene brachial plexus block was done Group U: ultrasound guided interscalene brachial plexus block was done Group NU: dual guidance (using both nerve stimulator and ultrasound) Group C: control group We assessed in each group: heart rate, noninvasive blood pressure, time needed for block, onset of sensory and motor power loss and their offset, and finally patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years old.
* Sex: Both sexes.
* ASA I & II.

Exclusion Criteria:

* - Patient refusal.
* Bleeding disorders.
* Damage or disease of the brachial plexus.
* ASA more than II.
* Pre-existing peripheral neuropathy.
* Patients with neuromuscular diseases.
* Patients with known hypersensitivity to drugs of the study.
* Patients with local skin infection at the site of injection.
* Psychiatric diseases interfering with evaluation of the block.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Analgesic effect of each technique | 12 hour
  using visual analogue scale for pain The patient is asked to express the degree of pain in numbers from 0-10, where 0 means no pain and 10 represents severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed K Mohamed, MD, Study Chair — Professor
Locations (1):
- Faculty of Medcine, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No